CLINICAL TRIAL: NCT04935476
Title: A Randomized, Placebo-Controlled, Multicenter Study to Assess the Safety and Efficacy of Dapsone for the Treatment of COVID-19 Positive Patients.
Brief Title: Dapsone Coronavirus SARS-CoV-2 Trial (DAP-CORONA) COVID-19
Acronym: DAP-CORONA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Pulmonem Inc. (Unknown)
Responsible Party: Principal Investigator, Jean Bourbeau, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PDC01
Record Dates: First submitted 2021-06-21; First posted 2021-06-23 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
Keywords: Dapsone; COVID-19; treatment for COVID-19; non-hospitalized patients; prophylaxis; SARS-COV-2; Clinical trials
MeSH Terms: conditions — COVID-19 | interventions — Dapsone; SDDS

STUDY DESIGN:
Intervention Model Description: This is a randomized, triple-blind, placebo-controlled, multi-center study.
  Following e-signature of the informed consent form, approximately 3000 participants meeting all inclusion criteria and no exclusion criteria will be randomized to receive either Dapsone or placebo (1:1 allocation ratio) for 21 days. Screening blood-work and confirmatory tests are made available to participants at their residence by the study. Study interventions (drugs or placebo) will be delivered directly to participants by courier .
  Participants are remotely followed-up through e-daily diary during 21 days of treatment along with virtual visits (phone) at 1, 7, 14, 21, 28 and 51 days following randomization for evaluation of the occurrence of any trial endpoints or other adverse events. During study enrollment patients are linked to the study through their participant account on the study virtual care platform.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, study staff and data analyst)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment (Active Comparator): Participants will receive standard of care and Dapsone per os (PO) twice daily for 21 days. If a dose is missed, it should not be replaced.
  Dosage form: Dapsone oral tablet
  Interventions: Drug: Dapsone 85 mg PO BID
- Control (Placebo Comparator): Participants will receive standard of care and placebo per os (PO) twice daily for 21 days. If a dose is missed, it should not be replaced.
  Dosage form: Placebo oral tablet
  Interventions: Drug: Placebo 85 mg PO BID

INTERVENTIONS:
Drug: Dapsone 85 mg PO BID — Participants will receive standard of care and study medication Dapsone 85 mg per os (PO) twice daily for 21 days. If a dose is missed, it will not be replaced.
  Other Names: diaminodiphenyl sulfone (DDS)
  Arms: Treatment
Drug: Placebo 85 mg PO BID — Placebo oral tablet, twice daily for 21 days.
  Other Names: Placebo
  Arms: Control

SUMMARY:
This is a multi-center, randomized, triple-blind, placebo-controlled (RCT) study to evaluate the efficacy and safety of Dapsone in older adults, and/or in adult patients (≥40yrs of age) with at least one high-risk comorbidity, among those with confirmed SARS-CoV-2 infection.

3000 infected patients diagnosed with COVID-19, non-hospitalized at the time of enrollment, meeting all inclusion and no exclusion criteria will be randomized (1:1 allocation ratio) to receive either Dapsone or placebo tablets for 21 days, and will be followed up for 7 days after treatment termination for outcome assessment and up to 30 days for safety monitoring.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether early treatment with Dapsone reduces pulmonary complications related to COVID-19 and consequent hospitalization in high-risk group of elderly adults and adults (≥40yrs of age) with comorbidity.

The secondary objectives are to determine the effect of Dapsone on reducing severe complications related to COVID-19 (ICU, intubation and death) and the safety of treatment with Dapsone in this high-risk COVID-19 patient population.

3000 patients will be enrolled to receive either Dapsone or placebo (1:1 allocation ratio) for 21 days. Follow-up assessments will occur remotely through participant e-daily diary and virtual visits (electronically via internet and/or telephone) at Day 1(start of study drug), 7, 14, 21, 28 and 51 following randomization in order to document the occurrence of any trial endpoints.

Safety and efficacy will be based on data from randomized patients. An independent data and safety monitoring committee (DSMC) will periodically review study results and will make recommendations to the study Steering Committee for continuing the trial as planned (or with modification) or for stopping early for safety concerns.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 40 years;
2. Symptomatic adults with confirmed COVID-19 (SARS-COV-2 PCR positive) for at least 24 hrs. and no more than 7 days: by report or observation, including one or more of the following: temperature ≥ 38°C (≥100.4°F), chills or shivering, cough, difficulty breathing, fatigue, headache, muscle or body ache, anosmia (loss of smell) and/or dysgeusia (loss of taste), GI symptoms (nausea and/or vomiting);

(3a) Aged ≥70 years or above, presence of concomitant comorbidity not required for inclusion

or

(3b) Aged ≥40 to <70 years, and presence of at least one of the following concomitant comorbidities by report, history, or observation:

* Cardiovascular diseases (e.g., hypertension, coronary artery diseases, congestive heart failure, symptomatic arrhythmia, transient brain ischemia, stroke)
* Chronic respiratory diseases (e.g., Chronic Obstructive Pulmonary Disease (COPD), asthma, pulmonary fibrosis)
* Obesity (BMI >30 kg/m^2)
* Type 2 Diabetes
* Cancer (participant reported: stable >6 months as per treating doctor/oncologist)
* Autoimmune diseases (T1D, RA, PA, MS, IBD, AD, SS, HT, SLE)

  (4) Participant is considered suitable for continued management in the out-patient setting.

  (5) Non-pregnant non-breastfeeding women of reproductive age group not planning pregnancy and/or adopting advised contraception during the study and for 3 months after the last dose of study medication.

Exclusion Criteria:

1. Unable to provide consent; diagnosis of dementia or other significant neurocognitive disorder;
2. Current hospitalization;
3. Patient requiring long term oxygen treatment of > 5 L O2/min because of a chronic lung condition at time of recruitment;
4. Known intolerance/allergy to sulfone;
5. Pregnant or breastfeeding women or is considering becoming pregnant during the study and for 3 months after the last dose of study medication;
6. Concurrent malignancy on systemic chemotherapy or immunotherapy;
7. Significantly impaired renal function within the past year reported by history and estimated glomerular filtration rate (eGFR) < 60 mL/min at screening
8. Severely underweight (≤ 40 kg)
9. G6PD deficiency (previous jaundice, jaundice with foods such as beans, or medication such as sulfa drugs, NSAIDs, quinolones, hydroxychloroquine or vitamin C), significant blood dyscrasia or anemia (Hb <12.0 g/dL in women and <13.0 g/dL in men; platelet count <50 x 10^9/L or < lower limit of normal at screening)
10. Impairment liver function [> 2 times the upper limit of normal (ULN) at screening at screening for AST, ALT, ALP, GGT, albumin or bilirubin), liver cirrhosis or hepatitis
11. Current use of folic acid antagonists (such as pyrimethamine), nitrofurantoin or primaquine
12. Currently taking oral dapsone for dermatological or other indications
13. Currently taking hydroxychloroquine or if have taken it within the last 6 months
14. Currently on any of the following medications: Aminolevulinic acid; Cladribine; Clozapine; Deferiprone; Prilocaine; Saquinavir; Sodium nitrite, Rifampin or St. John's wort
15. Received any of the following vaccines in the last 1 year : Cholera vaccine live; Typhoid vaccine, live; BCG (Bacillus Calmette and Guérin)
16. Currently taking any the following anticonvulsants : carbamazepine, phenytoin, levetiracetam and gabapentin
17. Currently participating in other interventional trials
18. Inability to provide contact details of caregiver/ next of kin to be contacted for study follow-up as participant's surrogate
19. Currently taking trimethoprim

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Composite outcome: All cause pre-hospitalization death or all-cause hospitalization | 30 days post randomization
  Number of participants requiring hospitalization or die prior to hospitalization in the first 30 days after randomization.

SECONDARY OUTCOMES:
Severe complications (composite outcome: All cause ICU admission, invasive ventilation or pre- or post-hospitalization death) | 30 days post randomization
  Number of participants developing severe complications and need ICU admission, invasive ventilation or die in the first 30 days.
All-cause ICU admission | 30 days post randomization
  Number of participants requiring ICU admission in the first 30 days after randomization.
Intubation with mechanical ventilation | 30 days post randomization
  Number of participants requiring intubation with mechanical ventilation in the first 30 days after randomization.
All-cause death | 30 days post randomization
  Number of participants who die in the first 30 days after randomization.
Hospitalization with all-cause requirement of supplemental oxygen | 30 days post randomization
  Number of participants requiring hospitalization with supplemental oxygen in the first 30 days after randomization.
Length of hospital stay among participants | 30 days post randomization
  Duration of hospitalization among study participants requiring hospitalization in the first 30 days after randomization.
Drug safety (Adverse Event (AE) and Serious Adverse Event (SAE)) for short term therapy in COVID-19 patients | 30 days post randomization
  Number of participants developing AE and SAE in the first 30 days post randomization.
Patient reported outcome (e.g. patient reported COVID-19 related symptoms) | 30 days post randomization
  Trajectory of participant reported COVID-19 related symptoms among study participants in the first 30 days after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bourbeau, MD,MSc,FRCPC, Principal Investigator — RI-MUHC
Locations (7):
- United States (5):
  - Arizona Pulmonary and Medical Specialists, Phoenix, Arizona
  - Peters Medical Research, LLC, High Point, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh UPMC, Pittsburgh, Pennsylvania
  - Principle Research Solutions, Spokane, Washington
- Canada (2):
  - Inspiration Research Limited, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No